CLINICAL TRIAL: NCT05601089
Title: Inter-Tester Reliability Of the Cumulated Ambulation Score in Patients With Stroke (InTRO-CAS-stroke)
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: University College Copenhagen (Other)
Responsible Party: Principal Investigator, Christian Hedelund Arens, Physiotherapist, MSc, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: P-2022-518
Record Dates: First submitted 2022-10-23; First posted 2022-11-01 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: Reliability; Cumulated Ambulation Score; Stroke; Inter-rater reliability; Inter-tester reliability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CAS is a measurement of basic mobility describing the degree of independence in three activities; getting in and out of bed, sit-to-stand from a chair with armrests, and indoor walking - each assessed on a three-point ordinal scale (0-2), resulting in a total one-day CAS between 0-6 points. Psychometric properties of the CAS has not been investigated i stroke. The design is an inter-tester reliability study.

DETAILED DESCRIPTION:
Rationale:

There are 12,000 new cases of stroke every year in Denmark. Stroke is the leading cause of adult disability, and more than 90,000 people are living with stroke. Many stroke survivors are in the need of help from others due to psychological, cognitive, physical, communication and/or swallowing problems. Stroke victims suffer from different impairments, resulting in different activity limitations. In Denmark, all stroke patients are admitted to a specialized acute stroke unit. The rehabilitation, if needed, is commenced within the first 48 hours of admission and continues throughout the hospital stay. In cases where patients need continued rehabilitation at discharge, then the municipality is advised where the rehabilitation continues.

At Copenhagen University Hospital Bispebjerg all patients receiving either physical or occupational therapy (or both) are tested with the Cumulated ambulation Score (CAS) as of 1st of April 2022. Each participant is tested at the beginning of the rehabilitation and before discharge. CAS is a measurement of basic mobility describing the degree of independence in three activities; getting in and out of bed, sit-to-stand from a chair with armrests, and indoor walking - each assessed on a three-point ordinal scale (0-2), resulting in a total one-day CAS between 0-6 points. CAS has shown to be reliable in both hip fracture and geriatric patients and useful in motoring basic mobility in geriatric patients. However, we do not know how reliable the score is in stroke victims. Therefore, the aim of this study is to investigate the inter-tester reliability of the three activities of the CAS and the total CAS.

Methods:

One experienced CAS user (NMJ) and one inexperienced (MM - last semester's physical therapy student) will be involved in the study. To achieve experience in using the CAS, the inexperienced CAS user will follow the experienced user throughout one day in regard to scoring the CAS. This will enable the inexperienced CAS user to get somewhat comfortable in the use of CAS.

Stroke victims experience changes in the basic mobility during the day, and even from hour to hour, due to spontaneous recovery, but also general tiredness and fatigue due to the brain damage can influence performances. Hence, the two therapists will only attend the patient at one session between day 1 and 4 after stroke onset, as soon as possible. Stroke victims will be tested after the instruction from one of the two raters randomly chosen by the random number generator software from GraphPad. Both therapists will be rating all three activities of the CAS on their own rating paper. The two raters will be blinded to each other's ratings until end of study, and hence not allowed to discuss their ratings before all participants has been assessed. A third person, not otherwise involved in scoring of patients, will collect, and hold the scoring cards directly after the ratings.

Furthermore, age, gender, premorbid disability level (premorbid Modified Rankin scale), height, weight, stroke severity (National Institute of Health - Stroke Scale, Scandinavian Stroke Scale), lesion type and localization will be collected of each stroke victim at baseline. Data from CAS at other timepoints, handgrip strength and 30 second sit-to-stand test will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic lesion relevant to this stroke event documented by CT/MRI
* NIHSS ≥ 2
* Patients eligible for physio- and/or occupational therapy planning

Exclusion Criteria:

- Not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult stroke survivors with the need for rehabilitation and a NIHSS-score of at least 2 at the Copenhagen University Hospital, Bispebjerg
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Inter-tester reliability of the Cumulated Ambulation Score | Tested by two raters once in a single session at day 1-4 after stroke onset (day of stroke = day 0). The study will end at completion of study or inclusion of all participants
  Agreement, percentage agreement, and linear weighted kappa between two CAS will be used for both the three activities independently and the total CAS-score to assess relative inter-tester reliability.
  Systematic between rater bias will be evaluated with the students t-test/Mann Whitney, as appropriate, and illustrated in a Bland Altman Plot. Furthermore, floor/ceiling of CAS sores will be assessed.
  Absolute reliability will assessed by intraclass correlation coefficient, standard error of the measurement SEM=SD×√(1-ICC) and the smallest real difference SRD=SEM×1.96×√(2)

CONTACTS AND LOCATIONS:
Overall Officials: Morten T. Kristensen, professor, Study Director — Department of Physio- and Occupational Therapy, Copenhagen University Hospital, Bispebjerg
Locations (1):
- Department of Physio- and Occupational Therapy, Bispebjerg, Copenhagen, Denmark

REFERENCES:
- [Derived] Arens CH, Johnsen NM, Milanesi M, Weli A, Linnebjerg C, Christensen H, Kristensen MT. Inter-tester reliability and agreement of the Cumulated Ambulation Score in acute stroke: The InTRO-CAS-stroke study. J Stroke Cerebrovasc Dis. 2024 May;33(5):107630. doi: 10.1016/j.jstrokecerebrovasdis.2024.107630. Epub 2024 Feb 5. PMID 38325673